CLINICAL TRIAL: NCT05410509
Title: "Embolization Before Ablation of Renal Cell Carcinoma (EMBARC)"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Principal Investigator, Andrew J. Gunn, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMBARC; 000536794 (Other Grant/Funding Number: Varian Medical Systems)
Record Dates: First submitted 2022-05-23; First posted 2022-06-08 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Renal Cell Carcinoma (RCC)
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RCC Participants (Experimental): Receive Trans-arterial embolization (TAE)
  Interventions: Procedure: Trans-arterial embolization (TAE)

INTERVENTIONS:
Procedure: Trans-arterial embolization (TAE) — Trans-arterial embolization (TAE) is a minimally-invasive procedure in which the tumor-feeding arteries are catheterized under x-ray guidance and therapeutically occluded. TAE of the kidney is routinely performed in clinical practice for traumatic or iatrogenic injury or to de-vascularize tumors such as angiomyolipomas, oncocytomas, and RCC. The procedure has a long clinical history of success with a very low major complication rate. TAE of RCC with or without percutaneous cryoablation (PA) has been described in retrospective case series as a mechanism to destroy the tumor, reduce bleeding complications from PA, or improve symptoms of RCC such as pain or hematuria. However, these findings have yet to be confirmed in a rigorous, prospective fashion.

SUMMARY:
Multi-center, single arm, prospective trial to estimate safety, feasibility, technical outcomes, and clinical outcomes of percutaneous cryoablation with neo-adjuvant trans-arterial embolization of the tumor in patients with T1b renal cell carcinoma. Continuous safety monitoring will be performed with stopping rules for patient accrual or study continuation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years
2. Solid renal mass consistent with RCC on either ultrasound, MRI, or CT
3. Longest tumor diameter measures 4.1-7cm
4. Tumor stage T1bN0M0 without vascular invasion, adenopathy, or distant metastatic disease
5. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to enrollment and agreement to use such a method during study participation
6. Provision of signed and dated informed consent form
7. Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

1. Pregnancy
2. Severe renal insufficiency with an Estimated Glomerular Filtration Rate (eGFR) <30
3. Renal cell carcinoma as part of a syndrome
4. Horseshoe kidney
5. Patient unable to undergo renal mass protocol CT or MRI
6. Severe allergy to iodinated contrast not mitigated by steroid and diphenhydramine prophylaxis
7. Uncorrectable coagulopathy, including a platelet count of <30,000/μL and/or an international normalized ratio (INR) >2.5 that does not respond to platelet transfusion or prothrombin complex concentrate infusion, respectively
8. Performance status precludes enrollment as determined by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of patients experiencing major adverse events defined as anything grade C or above by Society of Interventional Radiology Guidelines. | 30-90days post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Gunn, MD, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford Cancer Institute, Stanford, California
  - Mayo Clinic, Rochester, Minnesota
  - Thomas Jefferson Health, Philadelphia, Pennsylvania